CLINICAL TRIAL: NCT05658913
Title: Tau PET/CT Imaging in the Mismatch Prospective Cohort Study (MPC-TAU)
Acronym: MCP
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David Wolk, Principal Investigator, University of Pennsylvania
Other Study IDs: 850679
Record Dates: First submitted 2022-12-08; First posted 2022-12-21 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: AV-1451 — This is a cross-sectional study using the radiotracer AV-1451 to determine the relationship of tau pathology to other biomarker data of MPC participants.
  Other Names: 7-(6-[18F]fluoropyridin-3-yl)-5H-pyrido[4,3-b]indole

SUMMARY:
To collect Tau PET/CT imaging in older adults diagnosed with Mild Cognitive Impairment (MCI) or Alzheimer's Disease (AD) in the Mismatch Prospective Cohort Study (MPC-Tau) study to determine relationship to clinical, cognitive, and other biomarker data. Findings from this study will likely provide insight into the phenotypic variability of Alzheimer's Disease and other related pathologies.

DETAILED DESCRIPTION:
This is a cross-sectional study using the radiotracer AV-1451 to determine the relationship of tau pathology to other biomarker data of MPC participants. All subjects will already have been enrolled in the MPC Study. For the current protocol, participants will provide informed consent before beginning any study procedures. After screening assessments, participants will undergo PET/CT scan imaging with AV-1451.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in MPC study (Protocol 850160 at UPenn; Protocol 2022P002447 at MGH).
2. Reliable study partner to accompany participant to the PET/CT scan
3. A brain MRI must be performed within 6 months prior to their study AV-1451 TAU PET/CT scan date and be deemed of adequate quality that the scan may be used for study analysis, including 3T high-resolution imaging of medial temporal lobe structures.

Exclusion Criteria:

1. Have any medical or psychiatric conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study.
2. Have evidence of structural abnormalities such as major stroke or mass on MRI that is likely to interfere with analysis of the PET/CT scan.
3. Inability to tolerate or contraindication to imaging procedures in the opinion of an investigator or treating physician.
4. Have a history of significant ongoing alcohol or substance abuse based on self- report.
5. Female participants of child-bearing age will not be able to participate in this study, determined by self-report.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population includes individuals with a clinical diagnosis of MCI or possible/probably AD
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Clusters based on spatial pattern and extent of T-N Mismatch | 5 years
  We will test the hypotheses that spatial pattern and directionality of deviation in individual subjects of this metric will be correlated with modulatory factors such as non-AD pathology, brain resilience and vulnerability.
  Specifically, we will use hierarchical clustering to determine groups based on degree and spatial pattern of mismatch between tau PET and cortical thickness measured by MRI. In these groups, we will compare amount of white matter hyperintensities, degree of brain aging, and both cross-sectional and longitudinal cognitive measures, with the primary measure being the Clinical Dementia Rating scale sum of boxes.

CONTACTS AND LOCATIONS:
Overall Officials: David A. Wolk, Principal Investigator — University of Pennsylvania Department of Neurology at the Perelman School of Medicine; Sandhitsu R. Das, Principal Investigator — University of Pennsylvania Department of Neurology at the Perelman School of Medicine
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No